CLINICAL TRIAL: NCT07104955
Title: Single Cohort Before and After Mixed-methods Prospective Study to Investigate the Impact of the Salutare One Referral Software on Patient Outcomes, Safety and Effectiveness of Multi-Disciplinary Team (MDT) Meetings
Brief Title: Salutare One Referral Software Impact on Multi-Disciplinary Team (MDT) Meetings Effectiveness and Safety
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Salutare Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Salutare 01/2024; IRAS 347710 (Other: Health Research Authority)
Record Dates: First submitted 2025-06-18; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Cancer (Solid Tumors); Sarcoma
Keywords: digital health; digital health intervention; multi-disciplinary team meeting; MDT; digital health technology; referral; software
MeSH Terms: conditions — Neoplasms; Sarcoma

STUDY DESIGN:
Intervention Model Description: Prospective Before and After Study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- One Referral Group (Other): The study arm activities include:
  1. Pre-intervention phase: standard multi-disciplinary (MDT) process (without One Referral), baseline MDT meeting observation data collection, participants confirm informed consent and complete baseline survey.
  2. Onboarding phase: participants receive training on how to use the One Referral software and complete onboarding survey..
  3. Intervention phase: One Referral software is used as part of the MDT referral and review processes, MDT meeting observation data collection, participants complete intervention survey.
  4. Post-intervention phase: standard MDT process (without One Referral), follow-up MDT meeting observation data collection, participants complete offboarding survey
  Interventions: Other: MDT referral and review software

INTERVENTIONS:
Other: MDT referral and review software — Use of the multi-disciplinary team (MDT) meeting software to submit, review and discuss referrals

SUMMARY:
Multi-Disciplinary Team (MDT) meetings are crucial for planning patient care in the National Health Service (NHS), but they can be time-consuming and sometimes lack complete patient information. This can lead to delays in treatment decisions, potentially incomplete care plans, or the need to repeatedly discuss the same patient cases.

This study aims to test a new software called Salutare One Referral. One Referral is designed to make these meetings more efficient and effective. We want to see if this software can help healthcare staff prepare MDT referral information more easily and facilitate a more informed MDT discussion, which could lead to better patient care. If successful, this could help improve how MDTs operate across the NHS.

DETAILED DESCRIPTION:
This study aims to evaluate the safety, implementation effectiveness and feasibility of the Salutare One Referral software, a new tool designed to enhance Multi-Disciplinary Team (MDT) meetings. MDT meetings are recognized as the preferred means of delivering complex care for both chronic and acute diseases. However, there remains significant diversity in the purpose, structure, processes, and content of MDT meetings, as well as in how effectively they have been integrated into clinical practice.

Common issues observed in MDTs include:

* Deferring discussions due to incomplete medical history
* Re-discussing the same cases due to inadequate recording of previous discussions
* Failure to systematically manage cases to meet local and national targets The Salutare One Referral software is designed to address these challenges by streamlining the referral process, improving information sharing, and enhancing decision-making processes in MDT meetings. By potentially enhancing MDT efficiency, this study could lead to faster and better-coordinated patient care, reducing delays in treatment planning and implementation.

Study Design: This is a "before and after" study, observing MDT operations without the software, then with the software, followed by another period without it. MDT members will use the Salutare One Referral software during their regular meetings and complete questionnaires about their experience. The study will also analyse pseudonymized patient data to assess any changes in MDT review effectiveness. If successful, this study could lead to more efficient and effective MDT meetings, potentially resulting in improved patient care coordination across the NHS.

ELIGIBILITY:
Inclusion Criteria:

* MDT meeting Panel Members, Coordinators and staff submitting MDT referrals will take part in this study.

Exclusion Criteria:

* MDT meeting Panel Members, Coordinators and staff submitting MDT referrals who are unwilling or unable to take part in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-31 (Actual); Primary Completion 2026-06-19 (Estimated); Study Completion 2026-07-19 (Estimated)

PRIMARY OUTCOMES:
One Referral system safety in facilitating effective MDT meetings | 8 weeks (4 MDT meetings) for complex MDTs or 4 weeks (8 MDT meetings) for high-volume MDTs
  MDT panel participant feedback on safety and operational incidents
One Referral system implementation feasibility in facilitating effective MDT meetings | 8 weeks (4 MDT meetings) for complex MDTs or 4 weeks (8 MDT meetings) for high-volume MDTs
  MDT panel participant feedback on effectiveness (non-validated questionnaire)
One Referral system acceptability to MDT panel members acceptability in facilitating | 8 weeks (4 MDT meetings) for complex MDTs or 4 weeks (8 MDT meetings) for high-volume MDTs
  MDT panel participant feedback on acceptability (Software Usability Scale 0-100, higher score indicate a better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Moore, MD, Principal Investigator — Salutare Limited
Locations (1):
- Royal National Orthopaedic Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Participant consent provided for sharing de-identified data for the purpose of future research. Requests should be submitted to the sponsor and will be considered in line with the sponsor policy.

DOCUMENTS (1):
  • Study Protocol (2025-01-22): https://cdn.clinicaltrials.gov/large-docs/55/NCT07104955/Prot_000.pdf